CLINICAL TRIAL: NCT03213093
Title: Neurovascular Cutaneous Response to Pressure and Risk of Diabetic Foot Ulcer in Patients With Type 2 Diabetes
Brief Title: Pressure and Diabetic Foot
Acronym: PIV & MPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 69HCL16_0168
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Diabetes and Risk of Diabetic Foot Ulcer
Keywords: Diabetes; Diabetic Foot Ulcer; Plantar pressure
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diabetic patients with a risk of diabetic foot ulcer (Other)
  Interventions: Other: Measure of cutaneous microcirculation

INTERVENTIONS:
Other: Measure of cutaneous microcirculation — Measure of cutaneous microcirculation in response to a local application of pressure, to local heating and to the iontophoretic administration of acetylcholine

SUMMARY:
Diabetic foot ulcer (DFU) is a worldwide burden in the management of patients with diabetes. Peripheral neuropathy has a key role in the physiopathology of DFU. Others factors as skin vulnerability to plantar pressure, glycation of skin protein, articular rigidity, vascular component and abnormal foot plantar pressure are also important to take into account. The aim of the study is to assess prospectively different factors involved in DFU pathogenesis notably the neurovascular response to non noxious pressure.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Type 2 diabetic subject
* Absence of active diabetic foot ulcer
* Patients "Grade 0", "Grade 1", "Grade 2" or "Grade 3" of the International Working Group on Diabetic Foot Risk Classification defined by:
* absence of alteration of perception of Monofilament 10g at the level of the plantar arch for the "grade 0"
* alteration of perception of Monofilament 10g at the level of the plantar arch for the "grade 1"
* alteration of perception of Monofilament 10g at the level of the plantar arch associated with foot deformity and / or an arteriopathy defined by the absence of perception of one of the two peripheral pulses for the "grade 2"
* History of diabetic foot ulcer for the "grade 3"
* Signature of consent to participate in the study

Exclusion Criteria:

* Chronic alcoholism with usual consumption of at least 5 alcoholic drinks per day
* Pregnancy
* Congenital methemoglobinemia.
* Porphyria
* Skin injured on the tibia, whatever the lesion
* Recent major cardiovascular history (less than 3 months)
* Severe renal disease (serum creatinine> 300 μmol.l-1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
the rate of incidence of diabetic foot ulcer | At any time during a 3 years follow-up
  A diabetic foot ulcer is defined as a breakdown in the skin under malleolus

SECONDARY OUTCOMES:
Neurovascular response to pressure | At the end of the 3-year follow-up
  Receiver Operating Characteristic (ROC) analysis for neurovascular response to predict foot ulcer. Results are expressed in arbitrary unit.

CONTACTS AND LOCATIONS:
Locations (1):
- service d'endocrinologie, Centre Hospitalier Lyon Sud, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No